CLINICAL TRIAL: NCT03151590
Title: Non-Response to Exercise - Identification of Factors Contributing to Exercise Non-response.
Brief Title: Non-Response to Exercise
Acronym: NRE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Dr. Anja Boehm, Dr. med. (MD), University Hospital Tuebingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 446/2016BO2
Record Dates: First submitted 2017-05-09; First posted 2017-05-12 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Non-Responder
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: exercise training

SUMMARY:
The purpose of this prospective intervention study is to find biomarkers and underlying pathomechanisms for non-response of improvement in glucose metabolism to exercise.

An additional goal is to identify non-responders at an early stage, where prevention strategies (pharmacologically or by specific training) will be successful.

DETAILED DESCRIPTION:
At baseline and end of study, an intensive metabolic phenotyping including cerebral insulin sensitivity as well as tissue biopsies are performed in overweight untrained healthy participants at high risk for type 2 diabetes. During the study, an individual exercise training at 80% VO2max is performed for 9 weeks. Before and after the training intervention, acute tissue biopsies after a standardized bout of exercise are obtained.

ELIGIBILITY:
Inclusion Criteria:

* at least one of the following risk factors for type 2 diabetes:

  * overweight (BMI>27 kg/m2)
  * impaired fasting glucose and/ or glucose tolerance
  * former gestational diabetes
  * family history for type 2 diabetes (first-degree relative)
* sedentary participant (< 2 exercise bouts/week)

Exclusion Criteria:

* any kind of metal in or on the body
* thermosensory or heightened sensitivity to heating
* heightened sensitivity to loud noise or diseases of the ear
* claustrophobia
* Diabetes mellitus
* current pregnancy or breastfeeding
* cardiovascular diseases
* surgery, < 3 months ago
* participation in other clinical trials
* acute illness/infection, < 4 weeks ago
* severe mental illness
* hemoglobin, women < 11g/dl, men < 13g/dl
* potentially incompliant subjects and/or inability to absolve the exercise training
* glucose influencing drugs
* continuous analgetic drugs
* use of anticoagulants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
exercise response with respect to changes in insulin sensitivity from baseline to post-intervention measurement | 11 weeks
  insulin sensitivity is measured before and after the training intervention by a 5-point-75g-OGTT and calculated by ISI Matsuda

SECONDARY OUTCOMES:
molecular mechanisms of non-response | 11 weeks
  molecular mechanisms of non-response in insulin sensitivity in peripheral insulin target tissues (skeletal muscle, adipose tissue)
differences in the adaptation process to exercise in responders versus non-responders | 11 weeks
  by assessing the acute inflammatory response in blood samples and tissue biopsies obtained directly after an acute bout of exercise, at the beginning, and the end of the exercise intervention
inflammatory response to exercise | 11 weeks
  local (muscle and fat) versus systemic (blood) inflammatory response to exercise
changes in brain insulin sensitivity by exercise, and brain differences in responders vs. non-responders | 11 weeks
  changes in brain insulin sensitivity, before and after the intervention
role of visceral fat mass in determining the non-response of insulin sensitivity to exercise | 11 weeks
  measured by MRI
identification of serum biomarkers of non-response | 11 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Ulrich Häring, Prof., Study Director — University Hospital Tuebingen
Locations (1):
- Institute for Diabetes research and Metabolic Diseases of the Helmholtz Center Munich at the University of Tübingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kullmann S, Goj T, Veit R, Fritsche L, Wagner L, Schneeweiss P, Hoene M, Hoffmann C, Machann J, Niess A, Preissl H, Birkenfeld AL, Peter A, Haring HU, Fritsche A, Moller A, Weigert C, Heni M. Exercise restores brain insulin sensitivity in sedentary adults who are overweight and obese. JCI Insight. 2022 Sep 22;7(18):e161498. doi: 10.1172/jci.insight.161498. PMID 36134657
- [Derived] Hoffmann C, Schneeweiss P, Randrianarisoa E, Schnauder G, Kappler L, Machann J, Schick F, Fritsche A, Heni M, Birkenfeld A, Niess AM, Haring HU, Weigert C, Moller A. Response of Mitochondrial Respiration in Adipose Tissue and Muscle to 8 Weeks of Endurance Exercise in Obese Subjects. J Clin Endocrinol Metab. 2020 Nov 1;105(11):dgaa571. doi: 10.1210/clinem/dgaa571. PMID 32827042